CLINICAL TRIAL: NCT00040092
Title: A Study to Test the Effectiveness of Virulizin® Given in Combination With Standard Chemotherapy for Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aptose Biosciences Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOR/VIR/P03/002; NCT00045409 (obsolete NCT alias)
Record Dates: First submitted 2002-06-19; First posted 2002-06-20 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Pancreatic Cancer
Keywords: Virulizin; Immunotherapy; Pancreas; Pancreatic Cancer; clinical trial
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — virulizin

INTERVENTIONS:
Drug: Virulizin®

SUMMARY:
Virulizin is an immunotherapy drug preparation that is thought to stimulate the patient's immune system, which in turn may slow the growth of tumors. It is presented in vials as a sterile preparation for IM injection. The purpose of the trial is to investigate if Virulizin in combination with gemcitabine provides better efficacy than gemcitabine alone (with placebo) against pancreatic cancer.Virulizin® efficacy will continue to be assessed if chemotherapy is changed to 5-Fluorouracil.

DETAILED DESCRIPTION:
A Phase III, Double-blind, Multicenter, Randomized Study in Chemonaive Patients with Locally Advanced or Metastatic Pancreatic Cancer to Compare a Combination Therapy of Virulizin® plus Gemcitabine versus Placebo plus Gemcitabine; Optional Secondline Therapy may Include Continuation of Virulizin® or Placebo, Alone or in Combination with 5-Fluorouracil.

Patients who have not received any prior chemotherapy will be randomized to receive Gemcitabine plus Virulizin® versus Gemcitabine plus placebo in a double blind fashion. On disease progression patients may be switched to 5-Fluorouracil and continue to receive Virulizin® or placebo. Patients may continue Virulizin® alone, if clinically indicated when 5-Fluorouracil is discontinued.

ELIGIBILITY:
* Patients with advanced (unresectable or metastatic) pancreatic adenocarcinoma (TNM stages II, III or IV)
* No previous systemic chemotherapy(unless given as a radiosensitizer).
* ECOG Performance Status 0-2
* Life expectancy equal to or greater than 12 weeks
* Adequate laboratory and organ functions
* Stabilizable pain (stable analgesic intake)
* No radiotherapy during 4 weeks prior to trial entry
* No evidence of ascites, pleural effusion or third space fluid accumulation
* Not currently using, and have not used in 4 weeks prior to entering trial, systemic steroids or hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2002-07; Primary Completion 2005-07 (Actual)

REFERENCES:
- [Background] Ferdinandi ES, Braun DP, Liu C, Zee BC, Ely G. Virulizin(R) - A review of its antineoplastic activity. Expert Opin Investig Drugs. 1999 Oct;8(10):1721-1735. doi: 10.1517/13543784.8.10.1721. PMID 11139822
- [Background] Liu C, Ferdinandi ES, Ely G, Joshi SS. Virulizin-2gamma, a novel immunotherapeutic agent, in treatment of human pancreatic cancer xenografts. Int J Oncol. 2000 May;16(5):1015-20. doi: 10.3892/ijo.16.5.1015. PMID 10762639
- [Background] Warner E, Weinroth J, Chang S, MacDonald M, Strauss B. Phase II trial of Virulizin in patients with pancreatic cancer. Clin Invest Med. 1994 Feb;17(1):37-41. PMID 8174313